CLINICAL TRIAL: NCT02776774
Title: Topical Antibiotic Treatment for Spine Surgical Site Infection
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, David Flum, Director, Surgical Outcomes Research Center, University of Washington
Other Study IDs: STUDY00001775; 1R21AR068632-01 (NIH)
Record Dates: First submitted 2016-04-21; First posted 2016-05-18 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Surgical Wound Infection
Keywords: spine
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is considerable interest in using in-wound antibiotics (IWA) to prevent infection after spine surgery. An adequate evaluation of IWA is lacking and prior studies are limited by confounding and bias. This prospective study will enroll spine surgeons across the country to complete a survey about their knowledge, attitudes, and practices for using in-wound antibiotics.

DETAILED DESCRIPTION:
Surgical site infection (SSI) after spine surgery is a devastating complication. Spine SSIs occur in as many as 40,000 people each year, causing considerable disability and resulting in re-operative costs of over $100,000. Even with the use of standard perioperative infection prevention techniques, SSIs occur as often as 3-5% depending on the surveillance technique and time-window used, with widespread variability between practice sites and surgeons. A mainstay of SSI prevention is the timely administration of antibiotics, but one of the limits of intravenous antibiotic prophylaxis is that bone tissue concentrations of antibiotics are lower than blood levels. As a result, there has been increasing interest in the use of in-wound antibiotics (IWA), placed directly on the spine at the completion of surgery. IWAs have been supported by several observational studies with a recent systematic review suggesting an 84% decrease in SSI. However, most of these studies failed to address important confounding in the ways IWA were used and had variable follow-up. The only IWA randomized controlled trial (RCT), albeit underpowered failed to identify a protective effect, leading to uncertainty about the role of IWA. Because of the relative infrequency of SSI, variable windows of follow-up and high rates of confounding in prior studies of IWA a large scale trial of IWA with an appropriate follow-up period is needed to evaluate its effectiveness in spine surgery. Such a trial would be more feasible if randomization occurred at the level of hospital "cluster" (cRCT), to account for existing variation in practices regarding IWA use, variable rates of SSI, and use of other SSI prevention techniques.

Several pilot and feasibility questions need to be addressed before a cRCT of IWA can be proposed. SSI can appear as long as a year after spine surgery and short follow-up time in prior studies may have undercounted events and may have failed to recognize SSIs that may have been potentially delayed in detection because of the IWA. For example, the rationale for surgeon use of IWA, antibiotic type, or dose is unclear, as is whether surgeons use IWA in a similar fashion across patients and sites and if this represents confounding for which researchers must account. It is also unclear if surgeon use of IWAs is related to knowledge about existing data, beliefs and attitudes that may be barriers or enablers to a trial that promotes greater use of IWAs. To address these issues and direct an eventual cRCT, the investigators will perform surveys of spine surgeons assessing knowledge, behaviors and attitudes about IWA.

ELIGIBILITY:
Inclusion Criteria:

* Currently practicing spine surgeon, performing at least 5 spine surgeries per year
* Able to provide consent to participate in research
* 18 years of age or older

Exclusion Criteria:

* Surgeon or other provider that no longer performs spine surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spine surgeons across the United States
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Cizik, MPH, PhC, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-wound Antibiotics (IWA) Knowledge and Use: Compare knowledge, beliefs and attitudes about IWA with the actual use of IWA by surgeons.
Period: Overall Study
Arm/Group | Intra-wound Antibiotics (IWA) Knowledge and Use
Started (Total surveys submitted) | 91
Completed | 91 (Total after data cleaning)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Spine surgeons
Arm/Group | Intra-wound Antibiotics (IWA) Knowledge and Use
Number analyzed (Participants) | 91
Age, Customized [Count of Participants; unit: Participants] — Population: Age not captured in study
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex not captured in study
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Completed a clinical fellowship [Count of Participants; unit: Participants]
  Yes | 79
  No | 6
  Currently in fellowship | 3
  Missing | 3
Specialty [Count of Participants; unit: Participants]
  Neurological Surgery | 18
  Orthopaedic Surgery | 69
  Other | 1
  Missing | 3
Practice Type [Count of Participants; unit: Participants]
  Academic Center | 42
  Veterans Affairs Healthcare System | 0
  Physician Owned Group Practice | 15
  Community Health Center | 0
  Private Hospital | 10
  Solo/2 - Physician Practice | 6
  Group Practice, 3-5 | 4
  Group Practice, 6-50 | 6
  Group Practice, 50+ | 5
  Other | 0
  Missing | 3
Surgery Performance Location [Count of Participants; unit: Participants]
  Outpatient Surgery Center | 0
  Private Hospital | 37
  Public Hospital | 8
  Academic Center | 40
  Veterans Affairs Healthcare System | 0
  Other | 1
  Missing | 5
Opinion: Is IWA use for spine procedures the "standard of care"? [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Yes, for every spine procedure | 9
    Yes, but only for specific spine procedures | 36
    No | 46
Opinion: How often should IWA for spine procedures be used in practice? [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Routinely (75-100% of the time) | 29
    Selectively (<75% of the time) | 49
    Never | 3
    Don't know | 9
    Missing | 1
Opinion: The scientific evidence supporting the use of IWA is: [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Strong | 15
    Moderate | 44
    Weak | 26
    Evidence is non-existent | 0
    Don't know | 4
    Missing | 2
Opinion: Do IWA reduce the risk of infection by: [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    More than half | 31
    About half | 20
    Less than half | 16
    No benefit | 3
    Don't know | 20
    Missing | 1
Do you think a randomized trial on the use of IWA is needed? [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Yes | 71
    No | 19
    Missing | 1
Would you be willing to randomize your patients in a clinical trial on the use of IWA? [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Yes | 58
    No | 32
    Missing | 1
Do you use IWA in spine procedures for: [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    All patients | 14
    Some patients | 74
    No patients | 2
    Missing | 1
When did you first start using IWA? [Count of Participants; unit: Participants] — There was only one timepoint for this study (baseline). This variable was collected at the single timpoint and is not an outcome measure.
  Participants
    Less than 1 year ago | 5
    1-4 years ago | 49
    5 years ago or more | 34
    Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Attitudes About Using Intra-wound Antibiotics for Spine Surgery
Description: The investigators will compare answers to survey questions about knowledge of IWA among a diverse surgeon population to assess the feasibility of a future RCT and need for additional evidence.
Time Frame: Baseline
Population: Spine surgeon opinion regarding if intra-wound antibotic use for spine procedures is the "standard of care"?
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-wound Antibiotics (IWA) Knowledge and Use
Number analyzed (Participants) | 91
Participants
  Yes, for every spine procedure | 9
  Yes, but for only specific spine procedures | 36
  No | 46

2. Secondary Outcome: Describe Surgeon Practices for Using Intra-wound Antibiotics for Spine Surgery
Description: The investigators will survey surgeons about their current use of intra-wound antibiotics for spine surgery
Time Frame: Baseline
Population: Spine surgeons
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-wound Antibiotics (IWA) Knowledge and Use
Number analyzed (Participants) | 91
Participants
  Use, IWA on no instrumentation procedures: Never | 22
  Use, IWA on no instrumentation procedures: Sometimes | 46
  Use, IWA on no instrumentation procedures: Often | 6
  Use, IWA on no instrumentation procedures: Always | 12
  Use, IWA on no instrumentation procedures: Missing | 5
  Use, IWA on single level instrumentation procedure: Never | 5
  Use, IWA on single level instrumentation procedure: Sometimes | 31
  Use, IWA on single level instrumentation procedure: Often | 13
  Use, IWA on single level instrumentation procedure: Always | 37
  Use, IWA on single level instrumentation procedure: Missing | 5
  Use, IWA on multilevel instrumentation procedures: Never | 0
  Use, IWA on multilevel instrumentation procedures: Sometimes | 19
  Use, IWA on multilevel instrumentation procedures: Often | 18
  Use, IWA on multilevel instrumentation procedures: Always | 49
  Use, IWA on multilevel instrumentation procedures: Missing | 5

ADVERSE EVENTS:
Time Frame: Adverse Events not tracked and are inapplicable to this study.
Description: Adverse Events not tracked and are inapplicable to this study.
Arm/Group | Intra-wound Antibiotics (IWA) Knowledge and Use
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
It is unknown if participants that did not complete the survey would have been willing to participant in RCTs or not, or use IWA or not.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02776774/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02776774/SAP_001.pdf